CLINICAL TRIAL: NCT02047890
Title: An Open-label, Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics of BAY1000394 Given in a 3 Days on / 4 Days Off Schedule in Japanese Subjects With Advanced Malignancies
Brief Title: Japanese BAY1000394 Monotherapy Phase I Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15200
Record Dates: First submitted 2014-01-27; First posted 2014-01-28 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Neoplasms
Keywords: CDK inhibitor; BAY1000394; Advanced malignancies; Japanese
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY1000394 (Experimental): Approximately 12 subjects will be included: 3 to 6 evaluable subjects for each cohort. The cycle length will be 3 weeks (21 days).
  Interventions: Drug: BAY1000394 (2.5mg); Drug: BAY1000394 (5mg)

INTERVENTIONS:
Drug: BAY1000394 (2.5mg) — BAY1000934 2.5mg twice a day (bid) in a 3 days on and 4 days off schedule. (Cohort 1)
Drug: BAY1000394 (5mg) — BAY1000934 5mg twice a day (bid) in a 3 days on and 4 days off schedule. (Cohort 2)

SUMMARY:
This is an open-label, non-randomized, dose-escalating Phase I study to evaluate the safety, tolerability, pharmacokinetics of BAY1000394 given in a 3 days on / 4 days off schedule in Japanese subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female subjects aged ≥20 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
* Life expectancy of at least 12 weeks
* Subjects with advanced, histologically or cytologically confirmed solid tumors, not amenable to any standard therapy, have no standard therapy available, or subjects must have actively refused any treatment which would be regarded standard, and if in the judgment of the investigator, experimental treatment is clinically and ethically acceptable
* At least 1 tumor lesion evaluable by computer tomography (CT) or scan or magnetic resonance imaging (MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Adequate bone marrow, liver, and renal functions

Exclusion Criteria:

* Anticancer chemotherapy or immunotherapy within 4 weeks of study entry. Mitomycin C or nitrosoureas should not be given within 6 weeks of study entry.
* Radiotherapy to target lesions within 3 weeks prior to the first dose of study drug.
* Use of biological response modifiers, such as granulocyte colony-stimulating factor (G-CSF), within 3 weeks prior to the first dose of study drug.
* Symptomatic metastatic brain or meningeal tumors.
* Investigational drug treatment outside of this study during or within 4 weeks prior to study entry.
* Blood pressure <100/60 mmHg or pulse >100 BPM

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2018-07-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 6 months
Number of participants with abnormal lab parameters based on descriptive statistics | 6 months
Maximum observed drug concentration (Cmax) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose). Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Cmax divided by dose per body weight (Cmax,norm) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose). Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Cmax divided by dose (Cmax/D) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose). Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Area under the concentration versus time curve from zero to infinity after single dose (AUC) for BAY1000394 and its metabolite M-1 | = Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose)
AUC from time 0 to 12 hours after single dose (AUC(0-12) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8 and 12 hours
AUC divided by dose per body weight (AUCnorm) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose)
AUCnorm from time 0 to 12 hours after single dose (AUC(0-12),norm) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8 and 12 hours
AUC divided by dose (AUC/D) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose)
Time to reach Cmax (tmax) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose). Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Terminal half-life (t½) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 1: 0 (pre dose), 0.5, 1, 2, 4, 6, 8, 12 and 24 hours (Day 2, before morning dose). Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Maximum observed drug concentration after multiple dosing (Cmax,md) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Cmax divided by dose per body weight after multiple dosing (Cmax,norm,md) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
Cmax divided by dose (Cmax,md/D) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
AUC from time 0 to 12 hours after multiple dosing (AUC(0-12),md) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
AUCnorm from time 0 to 12 hours after multiple dosing (AUC(0-12),norm,md) for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)
AUC from time 0 to 12 hours divided by dose after multiple dosing for BAY1000394 and its metabolite M-1 | Cycle 1 / Day 10 : 0 (before morning dose), 0.5, 1, 2, 4, 6, 8 and 12 hours (before evening dose)

SECONDARY OUTCOMES:
Tumor response | Screening and on Day 21 of even numbered cycle

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Japan (2):
  - Kashiwa, Chiba
  - Fukuoka